CLINICAL TRIAL: NCT04747964
Title: A Phase 1,Multi-center, Randomized, Open, Single-dose Escalation Design to Evaluate the Safety, Tolerability and Pharmacodynamics of STSP-0601 for Injection in Patients With Inhibitory Hemophilia
Brief Title: A Safety Study of STSP-0601 in Adult Patients With Hemophilia A or B With Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STSP-0601-01
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-07

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A single lowest dose of treatment group (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- A single low dose of treatment group (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- A single low-intermediate dose of treatment group (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- A single intermediate dose of treatment group (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- A single high dose of treatment group (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- A single highest dose of treatment group (Experimental)
  Interventions: Drug: STSP-0601 for Injection

INTERVENTIONS:
Drug: STSP-0601 for Injection — Subjects will receive one single lowest dose of STSP-0601 for Injection following protocol requirements
  Arms: A single lowest dose of treatment group
Drug: STSP-0601 for Injection — Subjects will receive one single low dose of STSP-0601 for Injection following protocol requirements
  Arms: A single low dose of treatment group
Drug: STSP-0601 for Injection — Subjects will receive one single low-intermediate dose of STSP-0601 for Injection following protocol requirements
  Arms: A single low-intermediate dose of treatment group
Drug: STSP-0601 for Injection — Subjects will receive one single intermediate dose of STSP-0601 for Injection following protocol requirements
  Arms: A single intermediate dose of treatment group
Drug: STSP-0601 for Injection — Subjects will receive one single high dose of STSP-0601 for Injection following protocol requirements
  Arms: A single high dose of treatment group
Drug: STSP-0601 for Injection — Subjects will receive one single highest dose of STSP-0601 for Injection following protocol requirements
  Arms: A single highest dose of treatment group

SUMMARY:
This study will assess the pharmacokinetics and pharmacodynamics of STSP-0601 at six dose levels. The results will help identify the most optimal doses to treat bleedings in hemophilia patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤age≤65 years of age,male.
* Hemophilia A or B patients with inhibitors.
* Peak historical inhibitor titer ≥ 5 BU and a positive inhibitor test when enrolled.
* Establish proper venous access.
* Provide signed informed consent.

Exclusion Criteria:

* Have any coagulation disorder other than hemophilia A or B.
* Treat with prophylactic treatment of coagulation factor.
* Treat with anticoagulant within 7d of the time of study drug administration.
* Have an active, ongoing bleeding for which the patient is being treated, or treatment for a bleeding was stopped within 7d of the time of study drug administration.
* Have a history of arterial and/or venous thromboembolic events.
* Have platelet count <100,000/mL.
* Severe liver or kidney disease.
* Accept major operation or blood transfusion within 1 month of the time of screening.
* HIV antibody positive.
* Have a known allergy to Blood product.
* Participate in other clinical research within 1 month of the time of study drug administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects of adverse events | Baseline to Day 8
Number of subjects With Significant Abnormal Physical Examination | Baseline to Day 8
Number of subjects of Significant Abnormal Vital Signs Findings | Baseline to Day 8
Number of Participants With Significant Abnormal Laboratory Values | Baseline to Day 8
Number of subjects With Significant Abnormal Electrocardiography (ECG) Findings | Baseline,1 hour,4 hour,48 hour,Day 8

SECONDARY OUTCOMES:
Activated partial thromboplastin time | Baseline to 24 hours
Thrombin production (TG) peak | Baseline to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu W, Xue F, Fu R, Ding B, Li M, Sun T, Chen Y, Liu X, Ju M, Dai X, Wu Q, Zhou Z, Yu J, Wang X, Zhu Q, Zhou H, Yang R, Zhang L. Preclinical studies of a factor X activator and a phase 1 trial for hemophilia patients with inhibitors. J Thromb Haemost. 2023 Jun;21(6):1453-1465. doi: 10.1016/j.jtha.2023.01.040. Epub 2023 Feb 14. PMID 36796484